CLINICAL TRIAL: NCT02151175
Title: LIFUP for Treatment of Temporal Lobe Epilepsy
Brief Title: Low-intensity Focused Ultrasound Pulsation (LIFUP) for Treatment of Temporal Lobe Epilepsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: BrainSonix Inc. (Industry)
Collaborators: Gerald J. & Dorothy R. Friedman Center for Lymphedema Research & Treatment (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BX001
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy, Temporal Lobe
MeSH Terms: conditions — Epilepsy, Temporal Lobe

ARMS (1):
- LIFUP (Experimental)
  Interventions: Device: LIFUP

INTERVENTIONS:
Device: LIFUP

SUMMARY:
We intend to use focused ultrasound to stimulate or suppress brain activity in patients with epilepsy. We hypothesize that focused ultrasound is capable of brain stimulation or suppression visible with functional MRI, and will not cause tissue damage.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinical evidence from their diagnostic evaluations of unilateral hippocampal dysfunction and epileptogenicity.
* Subjects with seizures that have been refractory to treatment with at least three currently marketed antiepileptic drugs.
* Subjects with epilepsy who would clearly benefit from surgical intervention.
* Subjects who have been offered a non-dominant anterior-mesial temporal lobe resection as treatment for medication refractory epilepsy.

Exclusion Criteria:

* Subjects with a cognitive or psychiatric disorder that limits the ability to give informed consent or are unable to cooperate with the testing.
* Subjects with dementia, delirium and psychotic symptoms. - Subjects with ferromagnetic materials in the head.
* Subjects with severe cardiac disease, increased intracranial pressure, or a TENS unit.
* Subjects who exhibit primary generalized seizures or pseudoseizures.
* Subjects who have seizures secondary to drugs, alcohol, metabolic illness or progressive degenerative disease.
* Subjects who have experienced status epilepticus during the 3-week baseline period prior to the operation.
* Subjects (females) who are pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Absence of histological changes | 7 days

SECONDARY OUTCOMES:
Brief Symptom Inventory changes | 1 day
Beck Depression Inventory changes | 1 day
Neuropsychiatric changes | 1 day
Neurological changes | 1 day
Seizure frequency changes | 6 days

OTHER OUTCOMES:
Change in BOLD signal | Same day
Change in epileptiform discharges | Same day
Change in epileptiform discharge % | Same day

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Stern JM, Spivak NM, Becerra SA, Kuhn TP, Korb AS, Kronemyer D, Khanlou N, Reyes SD, Monti MM, Schnakers C, Walshaw P, Keselman I, Cohen MS, Yong W, Fried I, Jordan SE, Schafer ME, Engel J Jr, Bystritsky A. Safety of focused ultrasound neuromodulation in humans with temporal lobe epilepsy. Brain Stimul. 2021 Jul-Aug;14(4):1022-1031. doi: 10.1016/j.brs.2021.06.003. Epub 2021 Jun 23. PMID 34198105